CLINICAL TRIAL: NCT03525912
Title: Neuropsychiatric and Cardiovascular Side Effects in Ketamine Analgesic Infusions: a Prospective Study
Brief Title: Neuropsychiatric and Cardiovascular Side Effects in Ketamine Analgesic Infusions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Adriana Margarita Cadavid, Professor, Universidad de Antioquia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UdeA1002
Record Dates: First submitted 2018-04-21; First posted 2018-05-16 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Pain, Postoperative; Ketamine Adverse Reaction
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: single group assignment interventional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketamine infusion (Experimental): postoperative pain in adult population after abdominal, thoracic and orthopedic surgery that received adjuvant analgesia with ketamine 0.1mg/kg/h during 24 to 48 hours in postoperative period.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — continuous infusion of low dose ketamine for postoperative pain
  Other Names: analgesic ketamine

SUMMARY:
Evaluation of neuropsychiatric and cardiovascular side effects of low dose ketamine analgesic infusion for postoperative pain

DETAILED DESCRIPTION:
Postoperative pain is a world wide problem related with surgery. Multimodal analgesia may include ketamine, aimed to decrease opioid adverse effects in postoperative analgesia for major surgery, and risk of chronic postsurgical pain. Ketamine has shown efficacy as adjuvant in multimodal analgesia, however, neuropsychiatric and cardiovascular effects of ketamine at low doses in continue postoperative infusion are less known. This type of adverse effects may compromise appropriated recovery.

Objective

to determine frequency of delirium, agitation, sedation, hallucinations, bad dreams and cardiovascular changes associated with ketamine analgesic infusion treatment for postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

- patient scheduled for abdominal, thoracic or orthopedic surgery

Exclusion Criteria:

cognitive disfunction psychiatric illness cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Delirium | 2 days
  Presence or absence of delirium at 24 and 48 hours postoperatively over the past 2 days of exposure to ketamine infusion, using the Confusion Assessment Method (CAM), a clinical based assessment tool for identifying delirium. Consist of 4 criteria ( timing of symptoms, attention, thinking, consciousness). Considered to be positive for delirium if both features 1 and 2 are present, with at least one of features 3 or 4.

SECONDARY OUTCOMES:
Agitation | 24 and 48 hours postoperatively
  Richmond Agitation- Sedation Scale (RASS) score is a 10 point scale with discrete criteria, with four levels of agitation (+1 to +4), one level for calm and alert state (0), and 5 levels of sedation (-1 to -5)
Sedation | 24 and 48 hours postoperatively
  Clinician based Richmond Agitation- Sedation Scale (RASS) at 24 and 48 hours. RASS is a 10 point scale with discrete criteria, with four levels of agitation (+1 to +4), one level for calm and alert state (0), and 5 levels of sedation (-1 to -5)

OTHER OUTCOMES:
Hallucinations | 24 and 48 hours postoperatively
  Presence or absence of hallucinations
Bad Dreams | 24 and 48 hours postoperatively
  Presence or absence of bad dreams
Hypertension | 0, 24 and 48 hours postoperatively
  Hypertension is defined as a systolic blood pressure (SBP) of 140 mm Hg or more
Tachycardia | 0, 24 and 48 hours postoperatively
  a heart rate of more than 100 beats per minute (BPM)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana M Cadavid, MD, Principal Investigator — Anesthesiology professor
Locations (1):
- hospital universitario San Vicente Fundacion, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gorlin AW, Rosenfeld DM, Ramakrishna H. Intravenous sub-anesthetic ketamine for perioperative analgesia. J Anaesthesiol Clin Pharmacol. 2016 Apr-Jun;32(2):160-7. doi: 10.4103/0970-9185.182085. PMID 27275042
- [Background] Laskowski K, Stirling A, McKay WP, Lim HJ. A systematic review of intravenous ketamine for postoperative analgesia. Can J Anaesth. 2011 Oct;58(10):911-23. doi: 10.1007/s12630-011-9560-0. Epub 2011 Jul 20. PMID 21773855
- [Background] Li L, Vlisides PE. Ketamine: 50 Years of Modulating the Mind. Front Hum Neurosci. 2016 Nov 29;10:612. doi: 10.3389/fnhum.2016.00612. eCollection 2016. PMID 27965560